CLINICAL TRIAL: NCT03549208
Title: Single-blind, Single-center, Randomized, Active-controlled, Parallel Group, Phase I Study to Evaluate the Safety and Immunogenicity of Intramuscular Single Injection With Pneumococcal Conjugate Vaccine or Prevnar13 in Healthy Adults
Brief Title: A Study to Evaluate the Safety and Immunogeneicity of Multivalent Pneumococcal Conjugate Vaccine in Healthy Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LG-VECL003
Record Dates: First submitted 2018-05-25; First posted 2018-06-07 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-05

CONDITIONS: Pneumococcal Infection
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LBVE01 (Experimental): Multivalent pneumococcal conjugate vaccine
  Interventions: Biological: LBVE01
- LBVE02 (Experimental): Multivalent pneumococcal conjugate vaccine
  Interventions: Biological: LBVE02
- Prevnar13 (Active Comparator): Multivalent pneumococcal conjugate vaccine Prevnar13
  Interventions: Biological: Prevnar13

INTERVENTIONS:
Biological: LBVE01 — Multivalent pneumococcal conjugate vaccine be administered by Intramuscular injection into the thigh
  Arms: LBVE01
Biological: LBVE02 — Multivalent pneumococcal conjugate vaccine be administered by Intramuscular injection into the thigh
  Arms: LBVE02
Biological: Prevnar13 — 13-valent pneumococcal conjugate vaccine be administered by Intramuscular injection into the thigh
  Arms: Prevnar13

SUMMARY:
phase-1 study pneumococcal conjugate vaccine study in healthy adults

DETAILED DESCRIPTION:
A Study to Evaluate the Safety and Immunogeneicity of LBVE(Multivalent Pneumococcal Conjugate Vaccine) in Healthy adults

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult older than 19 years old and younger than 50 years old
* A subject who was informed of the purpose, method, and efficacy of the clinical study and signed the written informed consent form

Exclusion Criteria:

* A subject who participated in other clinical studies within 3 months before screening
* A subject who was vaccinated with other vaccines within 4 weeks before screening, or who is expected to receive other vaccination during the clinical study period
* A subject with medical history of hypersensitive reactions (e.g. anaphylaxis) to the test drug or its ingredients
* A subject who received immunoglobulin or blood-derived materials within 3 months before screening
* A subject with immunologic function disorders including congenital or acquired immunodeficiency disorders
* A subject who is receiving immunosuppressive therapy or drugs that can affect immunological reaction
* A subject with pyrexia of over 38 Celsius degrees on the day of the vaccination with the investigational products
* A subject with medical history of Invasive Pneumococcal Disease (IPD) or pneumonia caused by Streptococcus pneumoniae
* A subject who was vaccinated with any pneumococcal vaccine before screening
* A subject who received the vaccine containing diphtheria toxoid within 6 months before screening (e.g. adult Td vaccine)

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-07-25 (Estimated)

PRIMARY OUTCOMES:
Solicited adverse events | Baseline(pre-vaccination) up to 7 days after
  Solicited adverse events
Unsolicited adverse events | Baseline(pre-vaccination) up to 4 weeks after vaccination
  Unsolicited adverse events
Immediate reactions after vaccination | Baseline(pre-vaccination) up to 30 minutes after vaccination
  Immediate reactions after vaccination

SECONDARY OUTCOMES:
Serotype-Specific Pneumococcal immunoglobulin G antibody Geometric Mean Concentrations (GMCs) 4 weeks After Vaccination | 4 weeks After Vaccination
  GMC
Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) 4 weeks After Vaccination | 4 weeks After Vaccination
  GMT
Proportion of subjects achieving 4-fold rise in Pneumococcal Opsonophagocytic Activity (OPA) titer at 4 weeks after vaccination | 4 weeks after vaccination
  OPA titer

CONTACTS AND LOCATIONS:
Overall Officials: Myoung-don Oh, M.D., Principal Investigator — Seoul National University Hospital